CLINICAL TRIAL: NCT07093684
Title: Dementia and Kidney Disease: Epidemiological Approaches to Risk Factors and Treatment Strategies
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hong Xu, Assistant Professor, Karolinska Institutet
Other Study IDs: VR Starting grant #2022-01428
Record Dates: First submitted 2025-07-07; First posted 2025-07-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Acute Kidney Injuries; Real World Study; Dementia; Cholinergic System; Cognitive Decline; Alzheimer Dementia (AD); Cholinesterase Inhibitors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Swedish Dementia Registry (SveDem) Cohort: SveDem was established in 2007 with the purpose of increasing the quality of dementia care in Sweden. SveDem aims to register all dementia patients in Sweden at the time of dementia diagnosis and includes annual follow-ups. The registry stores data on demographics, living conditions, cognitive evaluation by Mini-Mental State Examination (MMSE), type of dementia, community support and pharmacological management.
  Interventions: Other: Kidney disease
- The SCREAM project: SCREAM is a healthcare utilization cohort of all Stockholm residents that accessed SLL healthcare and had a measurement of serum creatinine in either in- or outpatient care. The database includes 2 million individuals (and >60 million laboratory tests). The kidney function and other laboratory tests are already collected.

INTERVENTIONS:
Other: Kidney disease — This is a registry-based observational study investigating the association between kidney disease and dementia-related outcomes. Kidney disease is not assigned or manipulated by the researchers but is classified as an exposure based on diagnostic codes (e.g., ICD codes), and related laboratory test recorded in health registers.
  Groups: Swedish Dementia Registry (SveDem) Cohort

SUMMARY:
Kidney disease and dementia are both common in older adults, posing a significant burden on individuals and society. Growing evidence suggests that there may be links between the kidney and the brain. However, few studies have explored how these two conditions are connected in the general population. Understanding this link could help improve care for people living with either or both conditions.

This observational project aims to explore the two-way relationship between kidney disease and dementia. The main questions the investigators want to answer are:

1. Does kidney disease increase the risk or worsen the progression of dementia?
2. Does having dementia increase the risk or worsen the progression of kidney disease (both chronic and acute)?
3. Do reno-protective drugs help protect cognitive decline?
4. Do anti-dementia drugs help preserve kidney function?

To answer these questions, the investigators will analyze data collected over a period of 12 years, including people diagnosed with dementia, kidney disease, or both, using several large Swedish and international health registries:

1. The Swedish Dementia Registry (SveDem)
2. The Stockholm CREAtinine Measurements (SCREAM) project
3. The Swedish Renal Registry (SRR)
4. The GeroCovid Cohort
5. The Registry of Dementia of Girona (ReDeGi)
6. Cognitive impairment cohort from memory clinic, Karolinska University Hospital

This study will apply both traditional and advanced epidemiological methods, including multivariable regression, survival analysis, mixed-effects models, and machine learning (ML) techniques to examine long-term trends and associations.

ELIGIBILITY:
Inclusion Criteria:

* Population with dementia (all type) and kidney function measurements/Chronic kidney diagnosis

Exclusion Criteria:

* Population lack of important baseline and follow-up information such as year of birth and sex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project uses the Swedish Dementia Registry (SveDem), merged with the Stockholm CREAtinine Measurements (SCREAM) project, to access healthcare data and obtain measurements of serum creatinine from both inpatient and outpatient care. It also uses the Swedish National Patient Registry (NPR) to include diagnoses made in specialist clinics and hospitals, the Prescribed Drug Registry (which includes all prescribed medications), and the Total Population Register and Causes of Death Registry (CDR) to obtain dates of death.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Status Examination | MMSE will be assessed at baseline (dementia diagnosis) and at each follow-up visit every 12 months, up to 15 years or until death, whichever occurs first. Data will be reported at each time point and at study completion.
  The Mini-Mental State Examination (MMSE) is a standardized test used to screen for cognitive impairment and dementia. It assesses five domains of cognitive function including: orientation, registration, attention and calculation, recall, and language. The score range from 0 to 30. A score of 23 or lower is indicative of cognitive impairment. The MMSE takes only 5-10 minutes to test. MMSE is used at both baseline and follow-up visits.

SECONDARY OUTCOMES:
All-cause mortality | Will be assessed continuously from baseline up to 15 years until the end of follow-up.
  All-cause mortality will be defined as death from any cause, identified through linkage with the national death registry. Date of death will be recorded to calculate time-to-death from baseline.
Incidence of advanced dementia | Will be assessed annually from baseline (dementia) up to 15 years or until death, whichever occurs first.
  Advanced dementia will be defined based on MMSE score ≤10. MMSE scores range from 0 to 30, with lower scores indicating worse cognitive function. MMSE score will be identified from clinical follow-up records.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The data contains specific categories of personal data according to Article 9 of the General data protection regulation (GDPR) and KI is thus prohibited from sharing the data without an explicit consent from the registered or approval from the Swedish Ethical Review Authority (according to Section 3 and section 6 of the Ethical Review Act (2003:456)).

REFERENCES:
- [Background] Greenwald R. The handling of corneal donor tissue before penetrating keratoplasty. Todays OR Nurse. 1994 Sep-Oct;16(5):33-5. PMID 7974647
- [Background] Tsai HH, Yen RF, Lin CL, Kao CH. Increased risk of dementia in patients hospitalized with acute kidney injury: A nationwide population-based cohort study. PLoS One. 2017 Feb 13;12(2):e0171671. doi: 10.1371/journal.pone.0171671. eCollection 2017. PMID 28192452
- [Background] Xu H, Garcia-Ptacek S, Jonsson L, Wimo A, Nordstrom P, Eriksdotter M. Long-term Effects of Cholinesterase Inhibitors on Cognitive Decline and Mortality. Neurology. 2021 Apr 27;96(17):e2220-e2230. doi: 10.1212/WNL.0000000000011832. Epub 2021 Mar 19. PMID 33741639
- [Background] Saeed RW, Varma S, Peng-Nemeroff T, Sherry B, Balakhaneh D, Huston J, Tracey KJ, Al-Abed Y, Metz CN. Cholinergic stimulation blocks endothelial cell activation and leukocyte recruitment during inflammation. J Exp Med. 2005 Apr 4;201(7):1113-23. doi: 10.1084/jem.20040463. PMID 15809354
- [Background] Gansevoort RT, Correa-Rotter R, Hemmelgarn BR, Jafar TH, Heerspink HJ, Mann JF, Matsushita K, Wen CP. Chronic kidney disease and cardiovascular risk: epidemiology, mechanisms, and prevention. Lancet. 2013 Jul 27;382(9889):339-52. doi: 10.1016/S0140-6736(13)60595-4. Epub 2013 May 31. PMID 23727170
- [Background] Eckardt KU, Coresh J, Devuyst O, Johnson RJ, Kottgen A, Levey AS, Levin A. Evolving importance of kidney disease: from subspecialty to global health burden. Lancet. 2013 Jul 13;382(9887):158-69. doi: 10.1016/S0140-6736(13)60439-0. Epub 2013 May 31. PMID 23727165
- [Background] Wang J, Gu BJ, Masters CL, Wang YJ. A systemic view of Alzheimer disease - insights from amyloid-beta metabolism beyond the brain. Nat Rev Neurol. 2017 Sep 29;13(10):612-623. doi: 10.1038/nrneurol.2017.111. PMID 28960209